CLINICAL TRIAL: NCT04684849
Title: Assessment and Validation of Electronic Gas and Bloating Diary
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor of Medicine, Augusta University
Other Study IDs: 1541299
Record Dates: First submitted 2020-11-19; First posted 2020-12-28 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-07

CONDITIONS: Gas; Bloating; Distension; Constipation; Diarrhea
Keywords: Gas; Bloating; Distension; constipation; diarrhea
MeSH Terms: conditions — Mucopolysaccharidosis IV; Dilatation, Pathologic; Constipation; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Subjects who are healthy without disease
  Interventions: Other: APP Diary; Other: Paper Diary
- Gas and Bloating patients: Patients with symptoms of gas and bloating
  Interventions: Other: APP Diary; Other: Paper Diary

INTERVENTIONS:
Other: APP Diary — Subjects keep a multi- item electronic digital App survey of symptoms for 2 weeks
Other: Paper Diary — Subjects keep a multi-item paper survey of symptoms for 2 weeks

SUMMARY:
The investigator's goal is to improve the patient's compliance and accurate capture of patient reported gas and bloating symptoms, by utilizing a phone application that interactively records each gas and bloating event in addition to bowel events and other bowel symptoms. Such an electronic stool diary may relieve the burden of using a paper daily stool diary. The investigator will compare and validate the electronic gas and bloating diary with the paper gas and bloating diary.

DETAILED DESCRIPTION:
Gas-related symptoms (GRS) such as abdominal bloating, flatulence, and belching are some of the most common gastrointestinal complaints posed by the general population. These are hallmark symptoms in patients with functional gut disorders like irritable bowel syndrome but have also been linked to conditions such as gut hypersensitivity, altered gut microbiota and altered gut motility. The main issue with grasping the full impact of these symptoms on a patients' quality of life is that they are largely subjective and thus almost impossible to standardize. However, given their pervasiveness there is merit attempting to gauge their severity in as objective a manner as possible in order to track disease progress and response to treatment. GRS can be widely irregular and requiring patients to call into the office to answer questionnaires post treatment or keep handwritten logs to turn in later can lead to inaccurate data collection that can hinder accurate diagnosis and management. The ubiquitous nature of smartphones and user-friendly interfaces of electronic applications allow for information to be logged/accessed remotely and securely, each log would have their own time stamp and be recorded in an organized, consistent manner.

ELIGIBILITY:
Inclusion/Exclusion for gas and bloating subjects:

Inclusion:

1. Anyone 18 to 80 years of age, inclusive with gas-related symptoms (GRS) such as gas and bloating, plus any of the following: distension, diarrhea, and/ or abdominal discomfort.
2. Normal upper endoscopy, normal colonoscopy (<5 years) if patient is > 50 years of age, normal computerized abdominal tomography scan, or a normal right upper quadrant scan

Exclusion:

1. Women of childbearing age will be asked if they are pregnant, and a negative response will be sufficient. No pregnancy test will be performed.
2. History of previous GI surgeries (except for cholecystectomy, hysterectomy, and appendectomy)
3. Significant co-morbid medical conditions, including stroke, COPD( Chronic Obstructive Pulmonary Disease) and cancers (except for non-melanotic skin cancer)
4. Recent hospitalization within 30 days of enrollment in this study
5. Recent History (within 4 weeks) of antibiotic use
6. Recent History (within one week) of a colonoscopy or barium study

Inclusion/Exclusion for healthy subjects:

Inclusion:

1. Anyone 18 to 80 years of age, inclusive with no medical problems and a negative bowel disease screening questionnaire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone ages 18 to 80 years with constipation and gas and bloating symptoms.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of electronic APP diary information with paper form gas and bloating diary in healthy subjects | 2 weeks each
  The gas and bloating parameters recorded in the paper form gas bloating diary over 2 weeks will be correlated with the electronic APP gas and bloating diary parameters using Pearson correlation in healthy subjects
Correlation of electronic APP diary information with paper form gas and bloating diary in gas and bloating subjects | 2 weeks each
  The gas and bloating parameters recorded in the paper form gas and bloating diary over 2 weeks will be correlated with the electronic APP gas and bloating diary parameters using Pearson correlation in gas and bloating subjects

SECONDARY OUTCOMES:
Flatulence (Gas) | 2 weeks each
  Frequency, duration, and severity of flatulence will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating .
Abdominal distension | 2 weeks each
  Frequency, duration, and severity of abdominal distension will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating .
Bloating | 2 weeks each
  Frequency, duration, and severity of bloating will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating .
Abdominal Pain | 2 weeks each
  Frequency, duration, and severity of abdominal pain will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Belching | 2 weeks each
  Frequency, duration, and severity of belching will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Indigestion | 2 weeks
  Frequency, duration, and severity of indigestion will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Nausea | 2 weeks
  Frequency, duration, and severity of nausea will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Vomiting | 2 weeks
  Frequency and severity of vomiting will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Number of Bowel Movements | 2 weeks
  The number of Bowel Movements will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Constipation | 2 weeks
  Frequency, duration, and severity of constipation will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.
Diarrhea | 2 weeks
  Frequency and severity of diarrhea will be compared between the APP and gas and bloating diary and between healthy subjects and patients with gas and bloating.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States